CLINICAL TRIAL: NCT00763204
Title: A Phase I, Randomized, Observer-blind, Single-center, Vehicle- And Comparator-controlled, Initial Dose-ranging Study To Assess The Antipsoriatic Efficacy Of Different Concentrations Of An2728 Cream In A Psoriasis Plaque Test
Brief Title: A Phase I Study to Assess Novel Cream in a Psoriasis Plaque Test
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: AN2728-PSR-103; 2007-006600-37 (EudraCT Number); C3291022 (Other: Alias Study Number)
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Psoriasis
Keywords: Plaque Type Psoriasis; Topical
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): AN2728 Cream, 2%
  Interventions: Drug: AN2728 Cream, 2%
- 2 (Experimental): AN2728 Cream, 1%
  Interventions: Drug: AN2728 Cream, 1%
- 3 (Experimental): AN2728 Cream, 0.3%
  Interventions: Drug: AN2728 Cream, 0.3%
- 4 (Placebo Comparator): AN2728 Cream Vehicle
  Interventions: Drug: AN2728 Cream Vehicle
- 5 (Active Comparator): Betnesol®-V Creme (betamethasone 0.1 %)
  Interventions: Drug: Betnesol®-V Creme, 0.1%

INTERVENTIONS:
Drug: AN2728 Cream, 2%
  Arms: 1
Drug: AN2728 Cream, 1%
  Arms: 2
Drug: AN2728 Cream, 0.3%
  Arms: 3
Drug: AN2728 Cream Vehicle
  Arms: 4
Drug: Betnesol®-V Creme, 0.1%
  Other Names: betamethasone 0.1%
  Arms: 5

SUMMARY:
The purpose of this study is to investigate dose-response relationship, antipsoriatic efficacy and safety of different concentrations of topical formulations with AN2728 in subjects with psoriasis vulgaris.

DETAILED DESCRIPTION:
The study will be performed in 12 male subjects with stable psoriatic plaques. The study preparations and the comparator will be tested observer-blind. Treatments will be randomly assigned to the test fields. All subjects will receive all treatments, with intraindividual comparison of the treatments.

Altogether six test fields will be examined per subject (four active AN2728 creams of different concentrations: 2 %, 1 %, 0.3 %, 0.03 %, the active ingredient-free vehicle, and a marketed corticoid preparation). The test fields will be treated occlusively over a study period of 12 days. Topical application of approximately 200 uL of each assigned intervention is administered per treatment, for a total of 10 treatments over a 12-day treatment period.

ELIGIBILITY:
Inclusion Criteria:

* male subjects aged 18 years or older
* subjects with psoriasis vulgaris in a chronic stable phase and stable plaques with an area sufficient for five treatment fields
* the physical examination must be without disease findings unless the investigator considers an abnormality to be irrelevant to the outcome of the study
* written informed consent obtained

Exclusion Criteria:

* subjects with psoriasis guttata or pustular psoriasis
* subjects who require systemically acting medications for the treatment of psoriasis, which might counter or influence the study objectives, e.g. corticosteroids, cytostatics
* local treatment with antipsoriatics (like vitamin D, dithranol, glucocorticosteroids; except for salicyclic acid in vaseline) in the 4 weeks preceding and during the study; and any antipsoriatic treatment on the plaques (including corticosteroids, except for salicyclic acid) in the 8 weeks preceding and during the study.
* systemic treatment with antipsoriatics in the three months preceding and during the study
* treatment with systemic or locally acting medications which might counter or influence the study aim (e.g. MAO inhibitors, anti-epileptic drugs, anti-psychotic drugs) or medications which are known to provoke or aggravate psoriasis, e.g. Beta-blocker, antimalarial drugs and lithium drugs within two weeks before the beginning of the study and during the study.
* known allergic reactions to the active ingredients or other components of the study preparations or comparators
* blood pressure and heart rate outside the following allowed ranges: systolic blood pressure 80-160 mm Hg, diastolic blood pressure 60 - 100 mm Hg, heart rate 40-120 beats/min
* evidence of drug abuse
* UV-therapy within 4 weeks before beginning and during the study
* Symptoms of a clinically significant illness that may influenced the outcome of the study in the 4 weeks before and during the study
* participation in another clinical trial involving pharmaceutical products in the 4 weeks preceding and during the study
* in the opinion of the investigator or physician performing the initial examination the patient should not participate in the study, e.g. due to probable noncompliance or inability to understand the study and give adequately informed consent
* subject is institutionalized because of legal or regulatory order

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2008-02-29 (Actual); Primary Completion 2008-03-07 (Actual); Study Completion 2008-03-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of the active study preparations compared to the corresponding vehicle using differences in infiltrate thickness on study day 12. | Day 12

SECONDARY OUTCOMES:
Change in infiltrate thickness | Day 8
Sonographic measurements of infiltrate thickness | Day 8, Day 12
The AUC of the infiltrate thickness | Day 8, Day 12
Clinical assessment scores for assessment of efficacy | Day 8, Day 12

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Bioskin GmbH, Hamburg, Germany